CLINICAL TRIAL: NCT01055574
Title: Physical Capability Outcomes After Single-Level ProDisc-L Total Disc Replacement or Single-Level Anterior Lumbar Interbody Fusion: a Multi-Center Clinical Trial
Brief Title: Physical Capability Outcomes After Single-Level PD-L vs Single-Level ALIF: a Multi-Center Clinical Trial
Status: Terminated | Type: Observational
Why Stopped: Unanticipated study design flaw; PCO evaluator interrater reliability was not performed.
Sponsor: Gundersen Lutheran Medical Foundation (Other)
Collaborators: Synthes USA HQ, Inc. (Industry)
Responsible Party: Principal Investigator, Humbert (Drew) Sullivan, Chair, Department of Neurosurgery, Gundersen Lutheran Medical Foundation
Other Study IDs: 2-09-05-002; 20092359 (Other: Western Institutional Review Board (WIRB))
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Last update posted 2011-09-09 (Estimated); Status verified 2011-09

CONDITIONS: Physical Capability Outcomes
Keywords: lumbar disc arthroplasty; total disc replacement; ProDisc L; anterior lumbar interbody fusion; lumbar spine surgery outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ProDisc-L: Subjects who received single-level ProDisc-L total disc replacement prior to physical capability evaluations
- anterior lumbar interbody fusion (AILF): Subjects who received single-level anterior lumbar interbody fusion prior to physical capability evaluations

SUMMARY:
The purpose of this study is to compare the physical capability outcomes of patients who undergo single-level ProDisc-L disc replacement with those of patients who undergo stand-alone, single-level anterior lumbar interbody fusion (ALIF). This study will be the first multi-center clinical study to use clearly measurable outcomes from physical tests to compare the results of lumbar disc arthroplasty with disc fusion.

DETAILED DESCRIPTION:
Physical capability testing will be conducted once before surgery and at 6 months and 1 year after surgery. Physical capability testing assesses the ability to perform a number of common tasks: the distance a subject can walk comfortably in 6 minutes; the amount of weight a subject can lift, push, pull, and carry; and the ability to squat and work bending forward in the kneeling and standing positions. The results of this testing will be evaluated to determine whether the subject's physical capability meets the physical requirements of their job, based on their responses to a pre-study questionnaire. Each physical capability testing session will require from 1 to 1 ½ hours of the subject's time. Physical capability testing will be provided without charge.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients will meet the following criteria based on clinically appropriate criteria per standard of care at individual institutions which may include but are not limited to

* skeletally mature; BMI < 40
* suffered from low-back pain with or without leg pain for 6 months or longer
* no evidence of spinal deformity on plain radiograph
* no evidence of angular instability on flexion extension radiographs
* severe and incapacitating low-back pain, defined as a score of 40% or greater on the Oswestry Disability Questionnaire
* a single level of degenerative disc disease at L34, L45, or L5-S1 on magnetic resonance imaging (MRI) scan
* discography, if indicated, reproduces pain at the level of degeneration noted on the MRI scan and is negative for pain reproduction at adjacent levels
* bone mineral density T-Score by DEXA Scan >-1.0 for any skeletal region
* computed tomographic (CT) scan demonstrates the absence of pars defect at the index level
* CT scan demonstrates the absence of significant facet arthropathy at the index level
* considered reasonable candidates for surgery in regard to psychological factors as determined according to the standard of care at each participating center

Exclusion Criteria:

* active systemic infection
* evidence of alcoholism
* spondylolisthesis of greater than grade 1
* clinically significant lumbar spinal stenosis
* allergy to implant materials
* isolated radicular syndrome
* vertebral body compromised by trauma at the index level.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The target study population are those meeting all the FDA criteria for ProDisc-L. Patients with third-party coverage for ProDisc-L that received surgical implantation of this device will be in one group. Patients without third-party coverage for ProDisc-L that underwent stand-alone ALIF with a device that incorporates fixation of the superior vertebral body to the inferior vertebral body, and where an osteoinductive biologic agent is placed within the device will be in the other group.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2009-10; Primary Completion 2011-12 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Change in physical capability outcomes (6 minute walk; squats; light board game task standing bent forward /kneeling; floor-to-waist lift; horizontal lift; static push/pull force) | pre-op, at 6mo., and at 12mo.

SECONDARY OUTCOMES:
Oswestry Disability Index | pre-op, at 6mo., and at 12mo
EQ-5D Health Questionnaire | pre-op, at 6mo., and at 12mo.
Visual Analog Scale (VAS) scores for pain severity and frequency | pre-op, at 6mo., and at 12mo.
SF-36 scores for the 8 Domains | pre-op, at 6mo., and at 12mo.

CONTACTS AND LOCATIONS:
Overall Officials: Humbert (Drew) G Sullivan, MD, Principal Investigator — Gundersen Lutheran Health System, LaCrosse, WI; Jack E Zigler, MD, Principal Investigator — Texas Back Institute, Plano, TX; John G Devine, MD, Principal Investigator — Eisenhower Army Medical Center, Augusta, GA
Locations (6):
- United States (6):
  - University of Colorado Denver, Denver, Colorado
  - Christiana Spine Center, Newark, Delaware
  - Capital Regional Medical Center, Tallahassee, Florida
  - Orthopaedic Surgery Associates of Marquette, PC, Marquette, Michigan
  - Texas Back Institute, Plano, Texas
  - Gundersen Lutheran Health System, La Crosse, Wisconsin

REFERENCES:
- [Background] Kuslich SD, Ulstrom CL, Griffith SL, Ahern JW, Dowdle JD. The Bagby and Kuslich method of lumbar interbody fusion. History, techniques, and 2-year follow-up results of a United States prospective, multicenter trial. Spine (Phila Pa 1976). 1998 Jun 1;23(11):1267-78; discussion 1279. doi: 10.1097/00007632-199806010-00019. PMID 9636981
- [Background] Fairbank J, Frost H, Wilson-MacDonald J, Yu LM, Barker K, Collins R; Spine Stabilisation Trial Group. Randomised controlled trial to compare surgical stabilisation of the lumbar spine with an intensive rehabilitation programme for patients with chronic low back pain: the MRC spine stabilisation trial. BMJ. 2005 May 28;330(7502):1233. doi: 10.1136/bmj.38441.620417.8F. Epub 2005 May 23. PMID 15911537
- [Background] Bertagnoli R, Yue JJ, Shah RV, Nanieva R, Pfeiffer F, Fenk-Mayer A, Kershaw T, Husted DS. The treatment of disabling single-level lumbar discogenic low back pain with total disc arthroplasty utilizing the Prodisc prosthesis: a prospective study with 2-year minimum follow-up. Spine (Phila Pa 1976). 2005 Oct 1;30(19):2230-6. doi: 10.1097/01.brs.0000182217.87660.40. PMID 16205353
- [Background] Bao QB, Yuan HA. Prosthetic disc replacement: the future? Clin Orthop Relat Res. 2002 Jan;(394):139-45. doi: 10.1097/00003086-200201000-00016. PMID 11795725
- [Background] McAfee PC, Cunningham B, Holsapple G, Adams K, Blumenthal S, Guyer RD, Dmietriev A, Maxwell JH, Regan JJ, Isaza J. A prospective, randomized, multicenter Food and Drug Administration investigational device exemption study of lumbar total disc replacement with the CHARITE artificial disc versus lumbar fusion: part II: evaluation of radiographic outcomes and correlation of surgical technique accuracy with clinical outcomes. Spine (Phila Pa 1976). 2005 Jul 15;30(14):1576-83; discussion E388-90. doi: 10.1097/01.brs.0000170561.25636.1c. PMID 16025025
- [Background] Fritzell P, Hagg O, Wessberg P, Nordwall A; Swedish Lumbar Spine Study Group. 2001 Volvo Award Winner in Clinical Studies: Lumbar fusion versus nonsurgical treatment for chronic low back pain: a multicenter randomized controlled trial from the Swedish Lumbar Spine Study Group. Spine (Phila Pa 1976). 2001 Dec 1;26(23):2521-32; discussion 2532-4. doi: 10.1097/00007632-200112010-00002. PMID 11725230
- [Background] Brox JI, Sorensen R, Friis A, Nygaard O, Indahl A, Keller A, Ingebrigtsen T, Eriksen HR, Holm I, Koller AK, Riise R, Reikeras O. Randomized clinical trial of lumbar instrumented fusion and cognitive intervention and exercises in patients with chronic low back pain and disc degeneration. Spine (Phila Pa 1976). 2003 Sep 1;28(17):1913-21. doi: 10.1097/01.BRS.0000083234.62751.7A. PMID 12973134
- [Background] Blumenthal S, McAfee PC, Guyer RD, Hochschuler SH, Geisler FH, Holt RT, Garcia R Jr, Regan JJ, Ohnmeiss DD. A prospective, randomized, multicenter Food and Drug Administration investigational device exemptions study of lumbar total disc replacement with the CHARITE artificial disc versus lumbar fusion: part I: evaluation of clinical outcomes. Spine (Phila Pa 1976). 2005 Jul 15;30(14):1565-75; discussion E387-91. doi: 10.1097/01.brs.0000170587.32676.0e. PMID 16025024
- [Background] Zigler J, Delamarter R, Spivak JM, Linovitz RJ, Danielson GO 3rd, Haider TT, Cammisa F, Zuchermann J, Balderston R, Kitchel S, Foley K, Watkins R, Bradford D, Yue J, Yuan H, Herkowitz H, Geiger D, Bendo J, Peppers T, Sachs B, Girardi F, Kropf M, Goldstein J. Results of the prospective, randomized, multicenter Food and Drug Administration investigational device exemption study of the ProDisc-L total disc replacement versus circumferential fusion for the treatment of 1-level degenerative disc disease. Spine (Phila Pa 1976). 2007 May 15;32(11):1155-62; discussion 1163. doi: 10.1097/BRS.0b013e318054e377. PMID 17495770
- [Background] Chung SS, Lee CS, Kang CS. Lumbar total disc replacement using ProDisc II: a prospective study with a 2-year minimum follow-up. J Spinal Disord Tech. 2006 Aug;19(6):411-5. doi: 10.1097/00024720-200608000-00007. PMID 16891976
- [Background] Gillet P. The fate of the adjacent motion segments after lumbar fusion. J Spinal Disord Tech. 2003 Aug;16(4):338-45. doi: 10.1097/00024720-200308000-00005. PMID 12902949
- [Background] Gross DP, Battie MC. Reliability of safe maximum lifting determinations of a functional capacity evaluation. Phys Ther. 2002 Apr;82(4):364-71. PMID 11922852
- [Background] Reneman MF, Brouwer S, Meinema A, Dijkstra PU, Geertzen JH, Groothoff JW. Test-retest reliability of the Isernhagen Work Systems Functional Capacity Evaluation in healthy adults. J Occup Rehabil. 2004 Dec;14(4):295-305. doi: 10.1023/b:joor.0000047431.40598.47. PMID 15638259